CLINICAL TRIAL: NCT03310723
Title: A Comparison of Pre-oxygenation Techniques in Pregnant Patients Prior to a Cesarean Delivery - A Randomized Clinical Trial
Brief Title: Pre-Oxygenation Techniques in Pregnancy
Acronym: POP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Anthony Chau, Clinical Assistant Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H17-01996
Record Dates: First submitted 2017-10-04; First posted 2017-10-16 (Actual); Results first posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Preoxygenation
MeSH Terms: interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Face Mask Preoxygenation (Active Comparator): Tidal volume breathing for via a face mask set at 100% oxygen and a rate of 15L/min.
  Interventions: Device: Face Mask preoxygenation
- Optiflow Preoxygenation (Experimental): Tidal volume breathing with the OptiFlow system applied at 100% oxygen and a flow rate of 30-70L/min.
  Interventions: Device: OptiFlow preoxygenation

INTERVENTIONS:
Device: Face Mask preoxygenation — Standard face mask preoxygenation.
  Arms: Standard Face Mask Preoxygenation
Device: OptiFlow preoxygenation — Preoxygenation using transnasal humidified rapid insufflation ventilatory exchange (THRIVE).
  Other Names: THRIVE
  Arms: Optiflow Preoxygenation

SUMMARY:
A trial comparing outcomes of two pre-oxygenation techniques in obstetric patients.

DETAILED DESCRIPTION:
Pre-oxygenation is performed prior to general anesthesia to prevent hypoxia during airway management. It is typically performed using a standard tight-fitting face mask; however, recent advances in oxygenation have occurred through the use of trans-nasal oxygen delivery devices, such as OptiFlow. There is limited evidence of the use of OptiFlow in the pregnant patient, and as such, this study aims to show that OptiFlow is as effective at pre-oxygenation as a standard tight-fitting face-mask technique in the pregnant population.

ELIGIBILITY:
Inclusion Criteria:

* Healthy (American Society of Anesthesiologists class 1 or 2), pregnant patients ≥36 weeks gestation scheduled for elective Cesarean delivery under neuraxial anesthesia.

Exclusion Criteria:

* Comorbidities likely to alter outcome of respiration and gas exchange.
* Patients only able to breathe through their mouth.
* Patients who are in active labour.
* Patients unable to tolerate a face mask being held over their mouth and nose.
* Patients with a Body Mass Index ≥40kg/m2.
* Patients who are unable to give informed consent.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-11-10 (Actual); Primary Completion 2018-01-18 (Actual); Study Completion 2018-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anton Chau, MD MMSc, Principal Investigator — University of British Columbia
Locations (1):
- BC Women's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Face Mask Preoxygenation: Tidal volume breathing via a face mask set at 100% oxygen and a rate of 15L/min.
  Face Mask preoxygenation: Standard face mask preoxygenation.
Period: Overall Study
Arm/Group | Standard Face Mask Preoxygenation | Optiflow Preoxygenation
Started | 20 | 20
Completed (Discontinued) | 20 | 17
Not Completed | 0 | 3
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Protocol Violation | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Face Mask Preoxygenation | Optiflow Preoxygenation | Total
Number analyzed (Participants) | 20 | 17 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.8 (4.3) | 34.6 (5.3) | 34.7 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 17 | 37
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 20 | 17 | 37
Baseline end-tidal oxygen concentration (EtO2) [Mean (Standard Deviation); unit: Percentage units] | 15.9 (1.2) | 15.9 (1.5) | 15.9 (1.35)

OUTCOME MEASURES:

1. Primary Outcome: End Tidal Oxygen Concentration (ETO2) Following Tidal Volume Breathing Using Either Face Mask or OptiFlow
Description: Concentration of oxygen at the end of a breath following 3 minutes of tidal volume breathing using either face mask or OptiFlow
Time Frame: From baseline ETO2 concentration to the end of 3 minutes of tidal volume breathing
Measure: Median (Inter-Quartile Range); unit: Percentage units of end-tidal oxygen
Arm/Group | Standard Face Mask Preoxygenation | Optiflow Preoxygenation
Number analyzed (Participants) | 20 | 17
Percentage units of end-tidal oxygen | 91.0 [89.3 to 92.7] | 87.4 [85.5 to 89.2]

2. Secondary Outcome: End Tidal Oxygen Concentration (ETO2) Following Vital Capacity Breaths Using Either Face Mask or OptiFlow
Description: Concentration of oxygen at the end of a breath following 8 deep breaths using either face mask or OptiFlow
Time Frame: From baseline ETO2 concentration to the end of 8 vital capacity breaths (approximately 3 minutes)
Measure: Median (Inter-Quartile Range); unit: Percentage units
Arm/Group | Standard Face Mask Preoxygenation | Optiflow Preoxygenation
Number analyzed (Participants) | 20 | 17
Percentage units | 91.8 [90.1 to 93.4] | 85.9 [84.1 to 87.7]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during study procedures (i.e., from baseline measurements to end of pre-oxygenation at 3 minutes).
Arm/Group | Standard Face Mask Preoxygenation | Optiflow Preoxygenation
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-23): https://cdn.clinicaltrials.gov/large-docs/23/NCT03310723/Prot_SAP_000.pdf